CLINICAL TRIAL: NCT01136486
Title: The Role of Persistent Pain on Neuro Psychological Functioning and Community Integration in Traumatic Brain Injury
Brief Title: Pain in Traumatic Brain Injury - Basile, MD
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Rosemarie Basile, Neuropsychologist; Clinical Coordinator, Brain Injury Program, Northwell Health
Other Study IDs: 03-015
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Head Trauma
Keywords: head trauma; traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The observation through a chart review of persistent pain on neuro psychological functioning and how it applies to the community integration with patients that had suffered traumatic brain injury.

DETAILED DESCRIPTION:
This pilot study is designed and conducted over a one year period by the PI, who then solely carried out this study from recruitment, to patient testing, to data entry. Pain was assessed with the Visual Analog Scale and patients underwent a brief battery of tests that included assessment of neuropsychological functions, mood, anxiety and community functions.

ELIGIBILITY:
Inclusion Criteria:

* documented history of traumatic brain injury
* 18 years or older

Exclusion Criteria:

* younger than 18 years old
* cannot read and write English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: history of traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a documented history of head trauma ranging from mild to severe, with and without complaints of pain presented to Staten Island University Hospital over a 1 year period were considered for this study.
Groups:
- Treatment Arm: Pain was assessed with the Visual Analog Scale and patients underwent a brief battery of tests that included assessment of neuropsychological functions, mood, anxiety and community functions.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Level of Severity of TBI: Four categories based on pain severity (no pain, mild, moderate and severe pain).
Arm/Group | Level of Severity of TBI
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  African america | 12
  caucasian | 38
  Hispanic | 5
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pain Severity
Description: Pain was assessed on a scale for 1 (no pain) to 10 (severe) pain. This is observational study so participants were only seen at one time point, when they were referred to the neuropsychology service.
Time Frame: Referral
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Severity of Pain by Severity of Injury
Number analyzed (Participants) | 56
units on a scale | 7 (1.4)

ADVERSE EVENTS:
Description: Adverse events were not collected or assessed
Arm/Group | Severity of Pain by Severity of Injury
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes